CLINICAL TRIAL: NCT02408536
Title: Observational Retrospective Study on Treatment and Outcomes in Patients With Low-grade Serous Ovarian Cancer
Acronym: MITO 22
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: MITO 22
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Low-grade Serous Ovarian Carcinoma; Recurrent Invasive Borderline Serous Ovarian Cancer
Keywords: chemotherapy; hormone therapy; borderline; low-grade; serous ovarian cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival tissue tumor samples in paraffin blocks for evaluation of diagnosis and biomarkers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single cohort: Retrospective analysis of all patients diagnosed, from 01/01/2000 to 01/01/2014, with low-grade serous ovarian cancer or invasive recurrence after surgery for borderline serous carcinoma

SUMMARY:
The purpose of this study is to retrospectively evaluate treatments and outcomes of patients with low grade serous ovarian carcinomas in Italy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis low-grade serous ovarian carcinoma
* OR invasive recurrence after surgical resection of borderline serous ovarian carcinoma
* Availability of archival tumor specimen (paraffin embedded block) for central analysis and evaluation for mutations
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* High-grade serous, mucinous, endometrioid, or any other non-low-grade serous ovarian carcinoma
* Unavailability of archival tumor specimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed, from 01/01/2000 to 01/01/2014, with low-grade serous ovarian carcinoma or with invasive recurrence after surgery for borderline serous carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
risk of recurrence in patients with low-grade serous ovarian carcinoma | two years
number of patients with objective tumor response after receiving chemotherapy | 6 months
number of patients with objective tumor response after receiving hormone therapy | 6 months
number of patients with objective tumor response after receiving combination hormonal and chemotherapy | 6 months
progression free survival | 2 years
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, MD PhD, Principal Investigator — NCI Naples; Chiara Della Pepa, MD, Principal Investigator — NCI Naples; Francesco Perrone, MD PhD, Principal Investigator — NCI Naples
Locations (1):
- Istitute Nazionale Tumori - Fondazione G. Pascale, Napoli, Italy

REFERENCES:
- [Derived] Musacchio L, Califano D, Bartoletti M, Arenare L, Lorusso D, Losito NS, Cormio G, Greggi S, Raspagliesi F, Valabrega G, Salutari V, Pisano C, Spina A, Russo D, Del Sesto M, Canzonieri V, Ferrau F, Zannoni GF, Loizzi V, Ghizzoni V, Casanova C, Tuninetti V, Ducceschi M, Del Vecchio V, Scalone S, Priolo D, Perrone F, Scambia G, Pignata S. Clinical characteristics and molecular aspects of low-grade serous ovarian and peritoneal cancer: a multicenter, observational, retrospective analysis of MITO Group (MITO 22). Br J Cancer. 2022 Nov;127(8):1479-1486. doi: 10.1038/s41416-022-01897-1. Epub 2022 Jul 22. PMID 35869143